CLINICAL TRIAL: NCT00373841
Title: Genomic and Proteomic Analysis of Disease Progression in Idiopathic Pulmonary Fibrosis
Brief Title: Genomic and Proteomic Analysis of Disease Progression in Idiopathic Pulmonary Fibrosis (IPF)
Acronym: GAP
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kevin F. Gibson, Professor of Medicine, University of Pittsburgh
Other Study IDs: STUDY19040326
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Lung; Fibrosis; Idiopathic; Biomarkers; Genomics; Longitudinal
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples necessary to analyze disease progression in patient with idiopathic pulmonary fibrosis over a long period of time.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to identify genetic and biologic markers that may predict the loss of lung function due to idiopathic pulmonary fibrosis. The studies will compare genetic and biologic markers of samples to changes in symptoms. The ultimate goal is to predict if or when patients are likely to experience a rapid decline in lung function due to disease progression.

DETAILED DESCRIPTION:
People who are diagnosed with idiopathic pulmonary fibrosis are asked to participate in this study. The subject must be treated at the Dorothy P. and Richard P. Simmons Center for Interstitial Lung Disease. Subjects, if consented, are required to perform tests so that research data can be collected. At the initial visit, patients are subject to having a blood draw, pulmonary function testing, echocardiograms, and CT scans as well as completing several questionnaires designed to measure how the patient is feeling. Follow up visits are then scheduled in 3-4 month intervals. Every 3-4 months blood samples will be collected while every 6-8 months the questionnaires will administered. If the patient enters a stage of accelerated decline in lung function, a bronchoscopy will be performed to collect residual bronchoalveolar lavage fluid for testing. All of the results of clinical and laboratory testing will be placed into the subjects research file.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 or older
* Diagnosis of Idiopathic Pulmonary Fibrosis
* Treated at the Simmons Center

Exclusion Criteria:

* Other Lung Illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 and older who have been diagnosed with IPF and referred by a Simmons Center doctor.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2005-10; Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin F Gibson, MD, Principal Investigator — University of Pittsburgh - Dorothy P. and Richard P. Simmons Center for Interstitial Lung Disease
Locations (1):
- Michelle F MacPherson, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Chien JW, Richards TJ, Gibson KF, Zhang Y, Lindell KO, Shao L, Lyman SK, Adamkewicz JI, Smith V, Kaminski N, O'Riordan T. Serum lysyl oxidase-like 2 levels and idiopathic pulmonary fibrosis disease progression. Eur Respir J. 2014 May;43(5):1430-8. doi: 10.1183/09031936.00141013. Epub 2013 Oct 31. PMID 24177001
- See also: Homepage for the Dorothy P. and Richard P. Simmons Center for Interstitial Lung Disease — http://www.upmc.com/services/pulmonology/interstitial-lung-disease/